CLINICAL TRIAL: NCT06417684
Title: Comparison of Amitriptyline to Lifestyle Modification as Intervention for Vestibular Migraine
Acronym: RCTVM
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Richard A. Roberts, Ph.D., Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 240605
Record Dates: First submitted 2024-05-11; First posted 2024-05-16 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Vestibular Migraine
Keywords: vestibular
MeSH Terms: interventions — Amitriptyline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Amitriptyline (Active Comparator): amitriptyline, tablet, 25 mg, once daily, 90 days
  Interventions: Drug: Amitriptyline
- Lifestyle Modification (Active Comparator): Written and video instructions to help improve restful sleep, mealtime regularity, avoidance of dietary triggers, and exercise for 90 days.
  Interventions: Behavioral: Lifestyle Modification

INTERVENTIONS:
Drug: Amitriptyline — 25 mg prescribed to be taken once daily for 90 days each evening.
  Arms: Amitriptyline
Behavioral: Lifestyle Modification — Written and video instructions to instruct the participant to improve restful sleep, exercise, avoidance of dietary triggers, and mealtime regularity.
  Arms: Lifestyle Modification

SUMMARY:
Vestibular migraine (VM) is one of the most common causes of vertigo attacks, affecting 1 - 5% of people. People with vestibular migraine have lower quality of life compared to others and some may experience completely debilitating symptoms. Symptoms include vertigo, nausea, head motion-induced dizziness, unsteadiness, balance problems, and lightheadedness. There is evidence the medication amitriptyline in isolation and also our lifestyle modification intervention in isolation can each help reduce symptoms of dizziness and headache in patients with VM. However, these data are observational and subject to various types of bias. The purpose of the current investigation is to determine outcomes from each intervention using randomized allocation of participants diagnosed with VM into either the amitriptyline arm or the lifestyle modification arm. The investigators will measure for change in dizziness using the Dizziness Handicap Inventory (DHI) and for change in headache using the Headache Disability Inventory (HDI). For participants in the lifestyle modification arm, the investigators will also measure for change in lifestyle factor to determine improvement on those intervention factors. Measures will be obtained pre-intervention to establish baseline, at 30 days, 60 days, and 90 days. the investigators will also re-survey participants one year after initiation of intervention to determine adherence and status.

DETAILED DESCRIPTION:
1.0 Background

Vestibular migraine (VM) is one of the most common causes of vertigo attacks, affecting 1 - 5% of people. People with vestibular migraine have lower quality of life compared to others and some may experience completely debilitating symptoms. Symptoms include vertigo, nausea, head motion-induced dizziness, unsteadiness, balance problems, and lightheadedness. Most reports of vestibular migraine management have focused on treatment with medications; however, the investigators have shown that intervention with lifestyle modification is also effective.

1.1 Lifestyle Modification for Vestibular Migraine Our lifestyle modification intervention focuses on improving four factors: avoidance of dietary triggers, regulated mealtimes, restful sleep, and exercise. By controlling these factors that are often exacerbating for patients with VM, the investigators decrease the symptoms of dizziness and headache. In our studies, the investigators measure outcomes with two validated instruments, the dizziness handicap inventory (DHI) and the headache disability index (HDI). Using this approach, the investigators have found significant improvement within two weeks of starting the lifestyle modification intervention. Further, the investigators have seen that 44.7 - 59% of participants experienced significant improvement in dizziness within 30 days while 13.2 - 18.5% of patients experienced significant improvement in headache. The investigators have shown that 39% of participants experience significant reduction in dizziness and 18% in headache at 105 days of lifestyle modification intervention (Roberts et al, 2021). The investigators have even seen that 25% of participants continue to have significant benefit of lifestyle modification on dizziness at 371 days. Only 2.6 - 3.6 % of patients report worsened dizziness and no one has reported worse headache. The investigators were also able to determine that restful sleep was the modifiable factor most important for improvement when participant group data is evaluated. This lifestyle modification intervention appears effective and safe with long-term outcomes better than reported for oral preventive migraine medication which has adherence rates around 25% at six months and 14% at one year.

1.2 Amitriptyline for Vestibular Migraine Amitriptyline is a medication that is mentioned often as a preventive treatment for VM. This medication is a tricyclic antidepressant (TCA) that blocks the reuptake of both serotonin and norepinephrine neurotransmitters. This medication is considered more sedating and has greater anticholinergic properties than other TCAs. For depression, therapeutic action begins in 2 - 4 weeks. In a retrospective study, Salmito et al. (2017) reported significant improvement in vestibular symptoms and headache for 13 patients treated with amitriptyline 25 mg measured at three months. The authors also included lifestyle modification so this is not solely a medication mediated effect. Domínguez-Durán et al. (2020) used 10 mg of amitriptyline daily, one hour before sleeping, in 18 of their patients with VM. Two participants stopped or did not take the medication as directed. The authors reported significant improvement in dizziness and headache at the five-week follow-up appointment. 12 of the patients reported xerostomia and 11 daytime somnolence as side effects. Neither Salmito et al. nor Domínguez-Durán et al. used the DHI or HDI to measure outcome, making it more challenging to compare across studies. There are some known contraindications to use of amitriptyline including: history of significant mental health problems, pregnancy, cardiac, liver or renal co-morbidities as well as diabetes and glaucoma. Amitriptyline has also been shown to increase seizure activity in patients with epilepsy.

1.3 Randomized Controlled Trials Although VM is among the most common causes of dizziness and is the most common cause of episodic vertigo, the majority of studies investigation outcomes efficacy are observational in design. These studies typically show improvement for the intervention, but the inherent bias in that type of investigation is reduced with the use of randomized controlled trials (RCTs). The process of randomizing allocation of a participant to an intervention arm should balance observed and unobserved participant characteristics between groups and allow attribution of any differences in outcome to the study intervention. Although there are approximately five RCTs comparing various pharmacologic interventions for VM, there are none including amitriptyline and there are none using lifestyle modification without pharmacologic intervention.

2.0 Rationale and Specific Aims There is evidence that amitriptyline in isolation and also our lifestyle modification intervention in isolation can both help reduce symptoms of dizziness and headache in patients with VM. However, these data are observational and subject to various types of bias. The purpose of the current investigation is to determine outcomes from each intervention using randomized allocation of participants diagnosed with definite VM into either the amitriptyline arm or the lifestyle modification arm. The investigators will measure for change in dizziness using the DHI and for change in headache using the HDI. For participants in the lifestyle modification arm, the investigators will also measure for change in lifestyle factor to determine improvement on those intervention factors. Measures will be obtained pre-intervention to establish baseline, at 30 days, at 60 days, and at 90 days. The investigators will also re-survey participants one year after initiation of intervention to determine adherence and status.

The investigators hypothesize that amitriptyline and lifestyle modification intervention will improve symptoms of dizziness and headache similarly in patients with vestibular migraine measured at 60 days, but that the improvement will occur sooner (30 days) for participants in the lifestyle modification arm. Further, the investigators hypothesize there will be fewer reported side effects from participants in the lifestyle modification arm compared to participants in the amitriptyline arm.

Although VM is now recognized as a common cause of vertigo, there are few RCTs comparing efficacy of interventions and there are none comparing lifestyle modification to amitriptyline. Therefore, the results of the proposed investigation are intended to fill a critical void in our understanding of management of one of the most common causes of dizziness.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adults
* Diagnosed with Definite Vestibular Migraine
* Currently prescribed rescue medication for migraine is acceptable

Exclusion Criteria:

* Non-English speaking
* Diagnosed and undergoing treatment for active Definite Meniere's disease
* Already using amitriptyline
* Contraindicated for intervention with amitriptyline including:
* Patients with Hepatic Impairment
* Patients with Renal Impairment
* Pregnancy
* Breastfeeding
* Elderly Patients
* Allergy to amitriptyline
* Heart attack
* Used an MAO inhibitor in the past 14 days
* Used an "SSRI" antidepressant in the past 5 weeks
* Bipolar disorder (manic-depression) or schizophrenia
* Mental illness or psychosis
* Stroke
* Seizures
* Diabetes
* Glaucoma
* Problems with urination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Dizziness | Baseline DHI pre-intervention, 30, 60, 90 days and 1 year.
  We will measure for change in dizziness using the Dizziness Handicap Inventory (DHI)
Change in Headache | Baseline HDI pre-intervention, 30, 60, 90 days and 1 year.
  We will measure for change in headache using the Headache Disability Inventory Inventory (HDI)
Side Effects | 30, 60, 90 days and 1 year
  Participants will tabulate the rates of any reported side effects

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Roberts, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No